CLINICAL TRIAL: NCT02494830
Title: Comparative Bioavailability Study of Ketamine and Norketamine After Single Dose Administration of Ketamine 10, 20, 40 and 80 mg Prolonged Release Tablets in Fasting State and 5 mg Ketamine Solution for Infusion in 15 Healthy Subjects in Serum, Urine and Feces
Brief Title: Single Dose Administration of Ketamine 10, 20, 40 and 80 mg and 5 mg Solution for Infusion in 15 Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ketamine_03_2014
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Anesthetic Drugs
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ketamine 5 mg intravenous (Experimental)
  Interventions: Drug: Ketamine
- ketamine 10 mg oral (Experimental)
  Interventions: Drug: Ketamine
- ketamine 20 mg oral (Experimental)
  Interventions: Drug: Ketamine
- ketamine 40 mg oral (Experimental)
  Interventions: Drug: Ketamine
- ketamine 80 mg oral (Experimental)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Intravenous infusion of 5 mg ketamine solution, diluted in 240 ml 0.9% saline within 30 min under fasting conditions on study day 1 and oral administration of one prolonged release tablet ketamine together with 240 ml table water under fasting conditions with increased dose (10, 20, 40 and 80 mg) and at least 7 days wash-out between the study days

SUMMARY:
This study is designed for descriptive pharmacokinetic characterization of ketamine and norketamine in serum, urine and feces after oral single dose administration of a new developed prolonged release tablet formulation containing 10, 20, 40 and 80 mg ketamine under fasting conditions and for descriptive pharmacokinetic characterization of ketamine and norketamine in serum, urine and feces after intravenous single dose administration of 5 mg ketamine solution for infusion within 30 min

DETAILED DESCRIPTION:
Ketamine, a cyclohexanone derivative, is a non-barbiturate anesthetic agent which has been available in clinical practice for more than 40 years. Ketamine was first synthesized in 1962 and patented in Belgium in 1963. Ketamine, a potent non-competitive N-methyl-D-aspartate (NMDA) receptor antagonist, has a recognized unique therapeutic value in human and veterinary medicine as an anesthetic with analgesic properties. Ketamine is considered as one of the World Health Organisation (WHO) essential drugs for the management of refractory pain.

Ketamine is widely used for the induction and maintenance of general anesthesia, usually in combination with a sedative and if required a muscle relaxant. When used as an intravenous (i.v.) or intra-muscular (i.m.) injection, ketamine is best suited for short procedures. With additional doses, or by i.v. infusion, ketamine can be used for longer procedures. Due to its pharmacodynamic properties, important clinical applications are mainly brief diagnostic ones and surgical procedures in paediatric patients and ambulatory anesthesia, treatment of burn patients, obstetrics, and for the induction and maintenance of anesthesia in trauma victims, hypovolemic patients, patients with septic or cardiogenic shock, and patients with pulmonary diseases. Other uses include sedation in the intensive care setting, and analgesia particularly in emergency medicine as well as treatment of bronchospasm / asthma. However, the use of ketamine for humans in the EU is restricted to special indications, due to the occurrence of emergence reactions. Outside the EU, its ease of use gives ketamine a major advantage under difficult circumstances (developing countries and remote areas).

For therapeutic purposes, ketamine is usually administered intravenously (i.v.) or intramuscularly (i.m.). Its hydrochloride salt is marketed under many brand names such as Ketanest, Ketalar, or Ketaset. Ketamine is a chiral compound. While most marketed ketamine preparations are racemic mixtures of R-(-)-ketamine and S-(+)-ketamine (1:1), formulations containing only the enantiomer S-(+)-ketamine are also commercially available (e.g. Ketanest® S, Pfizer Pharma GmbH). S-(+)-ketamine is approximately four times more potent than R-(-)-ketamine and twice as potent as the racemic mixture.

It is well-known that ketamine exerts analgesic effects at subanesthetic doses. Therefore, during the past 15-20 years, ketamine has been used as an analgesic in a wide range of pain settings, including acute (e.g. post-operative pain, pain during dental procedures) and chronic pain (e.g. central or peripheral neuropathic pain, cancer pain) conditions.

Although the drug is only approved for intramuscular injection and intravenous injection or infusion, ketamine is frequently used via other routes of administration, such as subcutaneous (s.c.) injection or infusion, rectal, oral, intranasal, transdermal (patch), intrathecal or epidural administration. Considering that no oral formulation is approved, the marketed solution for injection/infusion or an extemporaneous preparation was used in clinical studies investigating the efficacy of orally administered ketamine. For clinical (off-label) use, the solution for injection/infusion is generally employed for oral treatment.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* sex: male or female
* ethnic origin: Caucasian
* body mass index: > 18.5 kg/m² and < 30 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which will be judged by the clinical investigator not to differ in a clinically relevant way from the normal state
* heart frequency between 50 and 90 bpm
* blood pressure between 140 and 100 systolic and 90 and 60 diastolic
* written informed consent

Exclusion Criteria:

* hepatic and renal diseases and/or pathological findings, which might interfere with pharmacokinetics of the study medication
* existing cardiovascular or haematological diseases and/or pathological findings, which might interfere with the drug's safety, tolerability and/or pharmacokinetics (e.g. tachycardia > 90 bpm, bradycardia < 50 bpm, ischemic heart disease like angina pectoris instabilis or myocardial infarction in the last 6 months, hypertension > 140/90 mm Hg)
* gastrointestinal diseases and/or pathological findings (e.g. stenoses), which might interfere with pharmacokinetics of the study medication
* hypersensitivity to the active ingredient ketamine or any of the excipients
* (pre-) eclampsia
* poor or untreated hyperthyreosis
* increased intracranial pressure
* glaucoma or perforating eye injury
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes (or equivalent) per day
* positive results in HIV, HBV or HCV screenings
* volunteers, who are on a diet, which could affect the pharmacokinetics of the drug
* heavy tea or coffee drinkers (more than 1L per day)
* lactation, pregnancy test positive or not performed or women of child-bearing age without safe contraception, as described on page 18, ch. 7.4.1. (Note for Guidance on Non-clinical Safety Studies for the Conduct of Human Clinical Trials for Pharmaceutical (CPMP/ICH/286/95 modifications))
* volunteers, suspected or known, not to follow instructions of the clinical investigators
* volunteers, who are unable to understand the written or verbal instructions, in particular regarding the risks and inconveniences, they will be exposed to, as a result of their participation in the study
* volunteers, liable to orthostatic dysregulation, fainting, or blackouts
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* less than 3 months after last blood donation
* intake of thyroid hormones or sympathomimetics
* any medication within 4 weeks prior to the intended first administration of the study medication, which might influence functions of the gastrointestinal tract (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists, proton pump inhibitors, anticholinergics)
* any other medication within two weeks prior to the first administration of the study medication, but at least 10-time the half-live of the respective drug (except oral contraceptives)
* intake of grapefruit containing food or beverages within 14 days prior to administration of the study medication
* intake of poppy seed containing food or beverages within 14 days prior to administration of the study medication
* known allergic reactions to the active ingredients used or to constituents of the study medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
bioavailability (F) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12 16, 24 36, 48, 60 h after study medication
  of ketamine

SECONDARY OUTCOMES:
area under the concentrations-time curve (AUC) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12 16, 24 36, 48, 60 h after study medication
  of ketamine and norketamine
maximum concentration (Cmax) of the concentrations-time curve | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12 16, 24 36, 48, 60 h after study medication
  of ketamine and norketamine
time point of maximum concentration (Tmax) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12 16, 24 36, 48, 60 h after study medication
  of ketamine and norketamine
terminal half-life (T1/2) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12 16, 24 36, 48, 60 h after study medication
  of ketamine and norketamine
volume of distribution at steady state (Vss) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 h after study medication
  of ketamine
renal clearance (CLR) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12 16, 24 36, 48, 60 and 72 h after study medication
  of ketamine
metabolic clearance (CLM) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 92 and 120 h after study medication
  of ketamine
intestinal clearance (CLintestinal) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 92 and 120 h after study medication
  of ketamine
mean residence time (MRT) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12 16, 24 36, 48, 60 h after study medication
  of ketamine
mean absorption time (MAT) | before and 10, 20, 30, 40, 50 min and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12 16, 24 36, 48, 60 h after study medication
  of ketamine

OTHER OUTCOMES:
cumulative excretion into urine (Ae,urine) | 24, 48, 72, 92 and 120 h after study medication
  of ketamine and norketamine
cumulative excretion into feces (Ae,feces) | 24, 48, 72, 92 and 120 h after study medication
  of ketamine and norketamine

CONTACTS AND LOCATIONS:
Overall Officials: Werner Siegmund, Prof, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany